CLINICAL TRIAL: NCT02609204
Title: NOVA™ PERG (Pattern Electroretinogram)and FERG (Flash Electroretinogram): Establishment of Reference Values for PERG and FERG Measurements
Brief Title: Normative Database for Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG)
Acronym: DIOPSYS-ND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Glaucoma Specialist, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-426E
Record Dates: First submitted 2015-08-07; First posted 2015-11-20 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma
Keywords: Pattern Electroretinogram (PERG); Flash Electroretinogram (FERG)
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy Controls (Experimental): Participants with normal eye exams and no history of eye diseases will best tested with Diopsys NOVA.
  Interventions: Diagnostic Test: Diopsys NOVA

INTERVENTIONS:
Diagnostic Test: Diopsys NOVA — Healthy Controls will have both eyes tested by the Diopsys NOVA machine using Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG) modules.
  Other Names: Diopsys-ND

SUMMARY:
The main goal of the study is to compile a normative database for the Neuro Optic Vision Assessment (NOVATM) Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG) modules. This normalization intends to be included in a probabilistic analysis protocol to allow NOVATM PERG/FERG users to identify patients with results outside the normal ranges.

DETAILED DESCRIPTION:
Investigators plan to enroll 50 subjects at Wills Eye Hospital without any eye diseases.

Participants will undergo a complete eye examination to determine eligibility, including visual acuity testing, intraocular pressure (IOP) in millimeters of mercury (mmHG), and visual field (VF) testing.

Participants will then be tested with Diopsys NOVA™ PERG & FERG systems. For both tests, two electrodes are placed on the skin underneath each eye below the eyelashes. Participants' skin will be cleaned before electrodes are placed. A small amount of gel will be placed on skin where electrodes are placed for testing. Electrical responses are recorded with electrodes in response to visual stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers age 18 years
* older with normal eye exam

Exclusion Criteria:

* spherical refraction outside + 5.0 Diopters and cylinder correction outside + 3.0 Diopters.
* IOP (intraocular pressure) ≥ 22 mm Hg (millimeters of mercury)
* history of any type of glaucoma in either eye.
* Intraocular surgery in study eye (except non-complicated cataract or refractive surgery performed more than 1 year before enrollment).
* Best corrected visual acuity worse than 20/40.
* Evidence of diabetic retinopathy, diabetic macular edema, or other vitreo-retinal disease in either eye.
* Evidence of optic nerve, macula and/or retinal nerve fiber layer abnormality in either eye.
* Evidence of reproducible (false positives, fixation losses and false negatives ≤ 25% with no observable testing artifacts).
* Standard Automatic Perimetry (SAP) abnormality in either eye, defined as Pattern Standard Deviation < 5% level, and/or abnormal Glaucoma Hemifield test result, and/or any other pattern of loss which is consistent with a neurologic and/or ocular disease.
* Current or recent (within the past 30 days) use of an agent (by any administering method) known to affect visual function.
* Inability to obtain reliable PERG/FERG (Pattern Electroretinogram/Flash Electroretinogram) results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Jay Katz, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: 51 Participants with normal eye exams and no history of eye diseases will best tested with Diopsys NOVA (Neuro Optic Vision Assessment).
  Diopsys NOVA: Healthy Controls will have both eyes tested by the Diopsys NOVA machine using Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG) modules.
Period: Overall Study
Arm/Group | Healthy Controls
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: 51 Participants with normal eye exams and no history of eye diseases will best tested with Diopsys NOVA.
  Diopsys NOVA: Healthy Controls will have both eyes tested by the Diopsys NOVA machine using Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG) modules.
Arm/Group | Healthy Controls
Number analyzed (Participants) | 51
Age, Continuous [Mean (Full Range); unit: years] | 53.3 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 18
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Flash Electroretinogram (FERG) Module Using Diopsys NOVA (Neuro Optic Vision Assessment) Amplitude
Description: Clinical data from participants with a normal eye examination to establish expected normal values of Flash Electroretinogram (FERG) photopic negative response (PhNR) amplitude in micro volts.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: micro volts
Arm/Group | Healthy Controls
Number analyzed (Participants) | 51
micro volts | -1.68 (0.78)

2. Primary Outcome: Flash Electroretinogram (FERG) Module Using Diopsys NOVA Latency
Description: Clinical data from participants with a normal eye examination to establish expected normal values of Flash Electroretinogram (FERG) photopic negative response (PhNR) latency in milliseconds.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Healthy Controls: 51 Participants with normal eye exams and no history of eye diseases will best tested with Diopsys NOVA.
  Diopsys NOVA: Healthy Controls will have both eyes tested by the Diopsys NOVA (Neuro Optic Vision Assessment) machine using Pattern Electroretinogram (PERG) and Flash Electroretinogram (FERG) modules.
Arm/Group | Healthy Controls
Number analyzed (Participants) | 51
milliseconds | 107.39 (10.22)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

LIMITATIONS AND CAVEATS:
All participants came from the same location.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No